CLINICAL TRIAL: NCT07102277
Title: Outcome of Laparoscopic Percutaneous Extra-peritoneal Closure of Internal Ring With or Without Peritoneal Cauterization
Brief Title: Laparoscopic Percutaneous Extra-peritoneal Closure of the Internal Ring With or Without Peritoneal Cauterization
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Shalaby, Associate Prof. Pediatric Surgery Unit, Faculty of Medicine, Tanta University, Egypt., Tanta University
Other Study IDs: REC 713
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Laparoscopic Percutaneous Extra-peritoneal Closure; Internal Ring; Peritoneal Cauterization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Percutaneous Internal Ring Suturing (PIRS) with peritoneal cauterization at the internal ring.
  Interventions: Procedure: Percutaneous Internal Ring Suturing (PIRS) with peritoneal cauterization
- Group B: Percutaneous Internal Ring Suturing (PIRS) without peritoneal cauterization.
  Interventions: Procedure: Percutaneous Internal Ring Suturing

INTERVENTIONS:
Procedure: Percutaneous Internal Ring Suturing (PIRS) with peritoneal cauterization — Percutaneous Internal Ring Suturing with peritoneal cauterization at the internal ring.
  Groups: Group A
Procedure: Percutaneous Internal Ring Suturing — Percutaneous Internal Ring Suturing (PIRS) without peritoneal cauterization.
  Groups: Group B

SUMMARY:
This research project aims to evaluate pediatric patients who underwent laparoscopic Percutaneous Internal Ring Suturing (PIRS) for inguinal hernia.

DETAILED DESCRIPTION:
Inguinal hernia repair is the most common procedure performed by pediatric surgery trainees. Open hernia repair (OH) is considered the gold standard approach for children; however, laparoscopic repair (LR) has recently emerged as an alternative option.

Laparoscopic percutaneous extraperitoneal closure of internal inguinal ring (Laparoscopic Percutaneous Internal Ring Suturing) (PIRS) is one of the plainest and most dependable operations for pediatric inguinal hernia.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (3 months to 12 years) with diagnosed inguinal hernia.
* Underwent Laparoscopic Percutaneous Internal Ring Suturing (PIRS).
* Clear documentation of whether cauterization was performed.
* At least 6 months of postoperative follow-up available.

Exclusion Criteria:

* Recurrent or complicated hernias (incarcerated/strangulated).
* Previous abdominal or pelvic surgery.
* Missing or incomplete surgical records.
* Less than 6 months of follow-up.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This is a retrospective comparative cohort study, evaluating pediatric patients who underwent Laparoscopic Percutaneous Internal Ring Suturing (PIRS) for inguinal hernia between [January 2023] and [December 2024].
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of recurrence | 1 year post-procedure
  Incidence of recurrence was recorded.

SECONDARY OUTCOMES:
Incidence of postoperative complications | 24 hours postoperatively
  Incidence of postoperative complications such as seroma, hematoma, hydrocele, and wound infection were recorded.
Degree of pain | 24 hours postoperatively
  Degree of pain was assessed using Face, Legs, Activity, Cry, Consolability scale (FLACC) in patients <7 years, or using the visual analog scale (VAS)(0 represents "no pain" while 10 represents "the worst pain imaginable") in patients≥7 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.